CLINICAL TRIAL: NCT00660803
Title: Retrospective Brazilian Study of Fulvestrant in Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Dendrix - Scientific Information Architecture (Unknown)
Responsible Party: Jose Eduardo Neves - Medical Science Director, AstraZeneca
Other Study IDs: NIS-OBR-FAS-2007/1
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: Advanced Breast Cancer; Hormone Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Postmenopausal women with hormone-receptor positive, advanced breast cancer who have failed at least one previous endocrine therapy and who have been treated at any one of the participating centres with fulvestrant.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant
  Other Names: Faslodex

SUMMARY:
Characterize the demographic and clinical features, as well as the main treatment results, among patients with advanced breast cancer treated with fulvestrant in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Positive HR or ER by immunohistochemistry
* Postmenopausal status at the time of treatment with fulvestrant
* Failure of at least one previous endocrine therapy before treatment with fulvestrant.

Exclusion Criteria:

* Patients who are still undergoing treatment with fulvestrant will not be eligible to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitals and primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Time to tumour progression
Objective response

SECONDARY OUTCOMES:
Duration of treatment with fulvestrant
Time and duration of response
Overall survival

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo